CLINICAL TRIAL: NCT02524236
Title: Studying the Dose Response of 50 and 100 IU of Botox A Toxin Injection in the Prostates of BPH Patients.
Brief Title: Effect of 50 and 100 IU Doses of Botox A Toxin Injection in BPH Patients.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelbary, MD, FEBU, Beni-Suef University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1 Urology
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH, OAB, Botox, dose response
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox 50 IU (Active Comparator): Intervention: Botox 50 IU vial will be reconstituted with saline 0.9% to a total volume of 5 ml. All patients will receive five injections of 1 mL of the BoNT-A solution, including two injections in each lateral lobe (one proximal and one distal) and one injection in the median lobe. The injection depth will be 7-10 mm.
  Botox injection in the prostate
  Interventions: Drug: Botox injection in the prostate
- Botox 100 IU (Active Comparator): Intervention: Botox 100 IU vial will be reconstituted with saline 0.9% to a total volume of 5 ml. All patients will receive five injections of 1 mL of the BoNT-A solution, including two injections in each lateral lobe (one proximal and one distal) and one injection in the median lobe. The injection depth will be 7-10 mm.
  Botox injection in the prostate
  Interventions: Drug: Botox injection in the prostate

INTERVENTIONS:
Drug: Botox injection in the prostate — transrectal access of prostatic injection
  Other Names: transrectal injection of the prostate

SUMMARY:
The primary objective of this study is to compare the efficacy and safety of a single injection of 50 U and 100 U doses of BoNT-A for the treatment of BPH-associated LUTS.

DETAILED DESCRIPTION:
Patients and method:

Men with symptomatic BPH will be invited to participate in this prospective study. Inclusion criteria will be an age of above 50 years, persistent moderate to severe LUTS as determined by International Prostatic Symptom Score (IPSS) >8, peak urinary flow rate of less than 12 mL/s, and an enlarged prostate gland on digital rectal examination. Exclusion criteria will be history of previous surgery for BPH, presence of urethral stenosis, urinary tract infection, prostate or bladder cancer, history of pelvic surgery or radiotherapy, neurological diseases, urinary retention and BPH-associated complications requiring surgical treatment including bladder stone, and bilateral hydronephrosis.

Subjects will undergo further evaluation before treatment, including urine analysis, serum creatinine, prostate-specific antigen (PSA), Trans rectal prostatic and Trans abdominal urinary tract sonography, uroflowmetry, and measurement of post-void residual volume (PVR) via abdominal ultrasonography.

Just before the injection procedure, patients will be randomized to receive either 50 U or 100 U of BoNT-A.

* Intervention All patients submitted for intervention will receive oral antibiotics (oral levofloxacin and flagyl 500 mg) 2 days before injection. Patients will be instructed to avoid taking anticoagulants, such as aspirin, for at least seven days prior to the procedure. An enema will be done two to four hours before the ultrasound to clean out the bowel.

Injection procedure: With the patient lying in lateral position, local anesthesia is performed with 20 mL of lidocaine 2% solution injected transrectally via transrectal ultrasound then wait for 10-minutes. The two different BoNT-A doses (50 U or 100 U) will be reconstituted with saline 0.9% to a total volume of 5 ml. All patients will receive five injections of 1 mL of the BoNT-A solution, including two injections in each lateral lobe (one proximal and one distal) and one injection in the median lobe. The injection depth will be 7-10 mm. After the procedure, patients will remain under observation until they are able to void spontaneously without hematuria. Oral levofloxacin (500 mg once a day) will be administered for five days.

Follow up:

Evaluation will be performed one week, 3 and 6 months after treatment. They will include a clinical assessment of LUTS with the IPSS score as well as measurement of peak urinary flow rate and post void residual volume. Serum PSA level and prostate volume will be assessed at the 6th month. The primary endpoint is improvement of IPSS scores (at least 30% improvement from baseline to 3 months IPSS and/or maximum urinary flow rate) and safety. The study will be stopped if 1) a life threatening, disabling or fatal event related to the BONT-A injection occurred, or 2) 40% or more of the participants report a moderate or severe side effect related to the botulinum toxin injection.

After 3 months, patients showing no improvement within 50 u group will be reinjected another dose of 100 u and then reevaluated after 3 months of reinjection.

Statistical Analysis:

Data will be expressed as means with standard deviations (SD) and range or absolute values and fractions. Intergroup changes from baseline of continuous variables will be analyzed with analysis of variance for repeated measurements. Intragroup comparisons will be performed using the Student's paired t-test. Fisher's test is used for categorical variables. A sample size of 17 in each group has 80% power to detect a difference between means of 3.00 (units in the IPSS score), at a two-tailed significance level of 0.05 or less.

ELIGIBILITY:
Inclusion Criteria:

* persistent moderate to severe LUTS as determined by International Prostatic Symptom Score (IPSS) >8.
* peak urinary flow rate of less than 12 mL/s.
* an enlarged prostate gland on digital rectal examination.

Exclusion Criteria:

* history of previous surgery for BPH.
* presence of urethral stenosis.
* urinary tract infection.
* prostate or bladder cancer.
* history of pelvic surgery or radiotherapy.
* neurological diseases.
* urinary retention.
* BPH-associated complications requiring surgical treatment including bladder stone, and bilateral hydronephrosis.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
IPSS score improvement | 3 months

SECONDARY OUTCOMES:
Urinary flow rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Abdelbary, md, Principal Investigator — Beni-Suef University
Locations (1):
- Beni - Suef University, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided